CLINICAL TRIAL: NCT07160062
Title: The Effect of Mandala Painting on Perioperative Psychological Well-Being, Emotional Self-Efficacy and Anxiety in Gynecologic Cancer Patients: A Randomized Controlled Study
Brief Title: Mandala Painting on Perioperative Psychological Well-Being,Emotional Self-Efficacy,Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assoc. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-SBB-0325
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mandala Painting; Gynecological Cancers; Psychological Well-being; Anxiety
Keywords: Emotional Self-Efficacy
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Mandala painting
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Mandala painting — Each mandala painting process took a total of 35 to 50 minutes, consisting of 30 to 40 minutes for mandala painting and drawing and 5 to 10 minutes for explaining the painted mandala.
  Arms: Intervention group

SUMMARY:
Aim: The aim of this study was to investigate the effect of mandala painting on psychological well-being, emotional self-efficacy, and anxiety in gynecological cancer patients during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:-

* 18 years of age or older,
* Diagnosed with any type or stage of gynecological cancer,
* In the perioperative period and scheduled for surgery,
* Willing to participate in this intervention,
* With written consent,
* Volunteering to participate in the study

Exclusion Criteria:

* Those with a serious physical or mental illness,
* Those with intellectual or cognitive impairment,
* Those with serious perioperative medical complications,
* Those who withdrew or dropped out of the study early,
* Those who were not willing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Emotional Self-Efficacy Scale | change from before implamentation patent and after 1st and 3rd days of practice
  The Turkish adaptation of the scale developed by Kirk, Shutte, and Hine was conducted by Totan, İkiz, and Karaca. The scale consists of 32 items and is based on a 5-point Likert scale (1-Strongly disagree, 7-Strongly agree).
Psychological Well-Being Scale | change from before implamentation patent and after 1st, and 3rd day of practice
  The scale was developed by Diener et al. to integrate and complement psychological well-being data and to measure social and psychological well-being. The Psychological Well-Being Scale was adapted into Turkish by Telef. The Cronbach's Alpha internal consistency coefficient obtained in the reliability study of the scale was calculated as .80. The Psychological Well-Being Scale consists of 8 items.
State Anxiety Scale | change from before implamentation patent and after 1st and 3rd days of practice
  The State and Trait Anxiety Scale, developed by Spielberger et al., was adapted into Turkish by Öner and Le Compte. It consists of two sections, each containing 20 questions. The questions in the State Anxiety Scale (SAS), which measures short-term anxiety arising from a temporary dangerous situation, are on a 4-point Likert scale (1: Not at all, 2: A little, 3: Very much, 4: Completely).

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)